CLINICAL TRIAL: NCT02048163
Title: A Comparison of the Effect of Intermittent and Continuous Infusion of Meropenem on the Prevalence of Nausea in Pediatric Cystic Fibrosis Patients
Brief Title: Intermittent Versus Continuous Infusion Meropenem in Cystic Fibrosis
Status: Withdrawn | Type: Observational
Why Stopped: No subjects enrolled
Sponsor: Dayton Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DCH 2013-034
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2015-01

CONDITIONS: Cystic Fibrosis
Keywords: Meropenem; Nausea; Pharmacokinetics
MeSH Terms: conditions — Cystic Fibrosis; Nausea

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Short infusion meropenem: Meropenem 20 mg/ml IV will be administered at a dose of 40 mg/kg (maximum 2,000 mg) every eight hours for 12 doses and will be infused over a 30 minute period. An equal volume of normal saline will be infused at the same time over four hours.
- Prolonged infusion meropenem: Meropenem 20 mg/ml IV will be administered at a dose of 40 mg/kg (maximum 2,000 mg) every eight hours for 12 doses and will be infused over a four hour period. An equal volume of normal saline will be infused at the same time over 30 minutes.

SUMMARY:
The purpose of this study is to compare the incidence of nausea and vomiting following short intermittent versus prolonged intermittent infusion of meropenem.

DETAILED DESCRIPTION:
1. To assess the number of episodes of emesis following both short and prolonged intermittent infusion of meropenem.
2. To assess the number of episodes of emesis corresponding to the peak serum concentration of meropenem.
3. To assess the number of episodes of emesis corresponding to the area under the meropenem serum concentration time curve.
4. To assess reported nausea, measured through administered dosages of anti-nausea medication, following both short and prolonged intermittent infusion of meropenem.
5. To assess reported nausea, measured through administered doses of anti-nausea medication, corresponding to peak concentrations of meropenem.
6. To assess reported nausea, measured through administered dosages of anti-nausea medication, corresponding to the area under the serum concentration time curve
7. To assess reported nausea, measured through patient-reported nausea measured using pictorial scales of severity of nausea in pediatric patients, following both short and prolonged intermittent infusion of meropenem.
8. To assess reported nausea, measured through patient-reported nausea measured using pictorial scales of severity corresponding to the peak serum concentrations of meropenem.
9. To assess reported nausea, measured through patient-reported nausea measured using pictorial scales of severity corresponding to the area under the meropenem serum concentration time curve.

ELIGIBILITY:
Inclusion Criteria:

1. Be an admitted patient at Dayton Children's Hospital.
2. Between 7 and 21 years of age.
3. Have a documented CF diagnosis with one or more of the following clinical features:

   1. Sweat chloride > 60 mEq/liter as determined by quantitative pilocarpine iontophoresis test (QPIT).
   2. Two mutations (well characterized) in the cystic fibrosis transmembrane conductive regulator (CTFR) gene.
   3. Abnormal nasal potential difference.
4. Based on Hankinson/NHanes III criteria, are able to elicit an FEV1 > 25% but with < 95% predicted value when admitted.
5. Sputum or throat swab specimen positive for P. aeruginosa and have a history of at least one additional sputum culture positive for P. aeruginosa within the last 12 months.
6. Are able to perform an acceptable spirometry session (defined as 3 acceptable or usable efforts per ATS/ERS criteria upon admission).
7. Have not smoked tobacco within 28 days prior to Visit 1 and agree not to smoke for the duration of the study.
8. Are able to and have given written informed consent (if they are adults) or assent in combination with consent of their legal representative(s) (if they are minors) in a manner approved by the Institutional Review Board.
9. Patient is experiencing symptoms of CF exacerbation of CF: with any 4 of the following 12 signs or symptoms:

   * Change in sputum;
   * New or increased hemoptysis;
   * Increased cough;
   * Increased dyspnea;
   * Malaise, fatigue or lethargy;
   * Temperature above 38°C;
   * Anorexia or weight loss;
   * Sinus pain or tenderness;
   * Change in sinus discharge;
   * Change in physical examination of the chest;
   * Decrease in pulmonary function by 10 percent or more from a previously recorded value;
   * Radiographic changes indicative of pulmonary infection.

Exclusion Criteria:

1. History of hypersensitivity or intolerance to meropenem.
2. History of hypersensitivity or intolerance to granisetron.
3. Are pregnant, breastfeeding, or unwilling to practice a highly effective method of birth control or abstinence during participation in the study.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female patients with cystic fibrosis ages 7 to 21 who are admitted to Dayton Children's Hospital and who will receive meropenem as part of their treatment regimen.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Compare indices of nausea following both prolonged intermittent and short intermittent infusions of meropenem | Nausea will be assessed while patient is receiving 4 days of prolonged intermittent infusion and 4 days of short intermittent infusion.
  Nausea indices will be measured for each treatment arm by averaging the doses of granisetron requested by each patient, the number of episodes of emesis, and the nausea faces scale scores recorded by patients.

SECONDARY OUTCOMES:
Compare pharmacokinetic data to indices of nausea. | Pharmacokinetic data will be obtained following the third, fourth, or fifth dose of meropenem administered during of each arm of the study. Peak serum concentration and area under the serum concentration time curve will be compared to nausea indices.
  Blood samples will be obtained at 0.5, 1.0 and 1.5 hours after the third, fourth or fifth meropenem dose on each arm of the study. Area under the serum concentration time curve and peak serum concentrations will be compared to each of the nausea indices.

CONTACTS AND LOCATIONS:
Overall Officials: Pat Christoff, PharmD, Principal Investigator — Dayton Children's Hospital
Locations (1):
- Dayton Children's Hospital, Dayton, Ohio, United States

REFERENCES:
- [Background] Prescott WA Jr, Gentile AE, Nagel JL, Pettit RS. Continuous-infusion antipseudomonal Beta-lactam therapy in patients with cystic fibrosis. P T. 2011 Nov;36(11):723-63. PMID 22346306
- [Background] Norrby SR, Gildon KM. Safety profile of meropenem: a review of nearly 5,000 patients treated with meropenem. Scand J Infect Dis. 1999;31(1):3-10. doi: 10.1080/00365549950161808. PMID 10381210
- [Background] Lodise TP, Lomaestro BM, Drusano GL; Society of Infectious Diseases Pharmacists. Application of antimicrobial pharmacodynamic concepts into clinical practice: focus on beta-lactam antibiotics: insights from the Society of Infectious Diseases Pharmacists. Pharmacotherapy. 2006 Sep;26(9):1320-32. doi: 10.1592/phco.26.9.1320. PMID 16945055
- [Background] Du X, Li C, Kuti JL, Nightingale CH, Nicolau DP. Population pharmacokinetics and pharmacodynamics of meropenem in pediatric patients. J Clin Pharmacol. 2006 Jan;46(1):69-75. doi: 10.1177/0091270005283283. PMID 16397286
- [Background] Legrand T, Chhun S, Rey E, Blanchet B, Zahar JR, Lanternier F, Pons G, Jullien V. Simultaneous determination of three carbapenem antibiotics in plasma by HPLC with ultraviolet detection. J Chromatogr B Analyt Technol Biomed Life Sci. 2008 Nov 15;875(2):551-6. doi: 10.1016/j.jchromb.2008.09.020. Epub 2008 Sep 25. PMID 18848512
- [Background] Blumer JL, Reed MD, Kearns GL, Jacobs RF, Gooch WM 3rd, Yogev R, Willims K, Ewing BJ. Sequential, single-dose pharmacokinetic evaluation of meropenem in hospitalized infants and children. Antimicrob Agents Chemother. 1995 Aug;39(8):1721-5. doi: 10.1128/AAC.39.8.1721. PMID 7486908